CLINICAL TRIAL: NCT01559857
Title: Pioglitazone Treatment for Insulin Resistant Patients With Mood Disorders
Brief Title: Pioglitazone in Patients With Mood Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Natalie Rasgon, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R21MH093948-01A1 (NIH); R21MH093948-01A1 (NIH)
Record Dates: First submitted 2012-03-16; First posted 2012-03-21 (Estimated); Results first posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-03

CONDITIONS: Major Depressive Disorder; Insulin Resistance
Keywords: Depression; Insulin resistance; Mood disorder
MeSH Terms: conditions — Depressive Disorder, Major; Insulin Resistance; Depression; Mood Disorders | interventions — Pioglitazone; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone (Active Comparator): 50% of participants will be allocated to 12 weeks of treatment with 30 mg/day of Pioglitazone.
  Interventions: Drug: Pioglitazone
- Sugar pill (Placebo Comparator): 50% of participants will be randomized to 12 weeks of treatment with placebo pill.
  Interventions: Drug: Sugar Pill

INTERVENTIONS:
Drug: Pioglitazone — 30mg once daily for 12 weeks
  Other Names: Actos
  Arms: Pioglitazone
Drug: Sugar Pill — Placebo
  Other Names: Placebo
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to see how an insulin sensitizing medication, Pioglitazone, can cause changes in mood in some depressed patients. Study participants receive assessment of their cognitive and metabolic functioning.

If they meet criteria, they will be asked to take either Pioglitazone or a placebo for a 90-day trial. Participants will undergo an Oral Glucose Tolerance Test to measure fasting insulin and glucose levels, as well as routine blood testing.

The investigators hope to quantify the role of Pioglitazone in patients with mood disorders and compare the values to those previously obtained in a healthy age-matched control population. The investigators also hope to examine the association between IR and cognitive performance and clinical course of depression in patients with mood disorders.

DETAILED DESCRIPTION:
While the association between insulin resistance (IR) and depressive symptoms is well documented (Gold et al., 2005), causal aspects of the relationship are incompletely documented and likely bidirectional. As the current prevalence rates of DM2 and related diseases grow worldwide and its associated metabolic consequences become more salient, it is increasingly critical to understand the role of IR in depressive disorders.

Insulin has been shown to alter central nervous system (CNS) concentrations of neurotransmitters such as dopamine (Lozovsky et al., 1981) and norepinephrine (Boyd et al., 1985), by a variety of mechanisms, as well as to have direct electrophysiological effects on neuronal activity (Boyd et al., 1985). Additionally, induced IR in the CNS has been shown to result in cognitive and behavioral alterations in animal models (Kovacs and Hajnal, 2009).

Accordingly, when depression manifests as a sequela of metabolic disorders such as obesity and DM2, it is hypothesized to be associated with resistance of CNS structures to the effects of insulin, which may derive from genetic polymorphisms, as well as from long-term exposure to excess amounts of circulating insulin due to peripheral IR (Okamura et al., 2000b). Thus, "overcoming" central IR," for example by pharmacological interventions, could be an attractive strategy in the treatment and prevention of these disorders.

This study aimed to assess mood effects in a 12-week double-blind, randomized-controlled trial of adjuvant treatment with the PPARγ-agonist pioglitazone, an insulin-sensitizing agent, compared with treatment with placebo, in participants with non-psychotic, non-remitting depression receiving standard psychiatric regimens for unipolar or bipolar depression. Pioglitazone is an FDA-approved, insulin-sensitizing treatment for DM2 and has particularly beneficial effects on lipid profile (Goldberg et al., 2005) and rate of cardiovascular events (Lincoff et al., 2007) in this population. Furthermore, in assessing the utility of an additive insulin-sensitizing agent on mood outcomes in both insulin sensitive and insulin resistant patients, this study attempted to disentangle the role of insulin-sensitizing and anti-inflammatory mechanisms.

In an a prior manner, this study's aims were twofold: (1) to assess whether treatment with pioglitazone would result in significantly greater mood improvement compared to treatment with placebo among patients with unremitted depression despite treatment as usual (TAU) and (2) to examine mechanisms of proposed effects of a PPARγ-agonist on mood outcomes by comparing treatment outcomes based on surrogate markers of glucose metabolic status (hereafter referred to IR and IS) between IR and insulin sensitive (IS) participants.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 65 years
* BMI between 25 and 35
* Diagnosis of unipolar, non-psychotic, non-melancholic major depressive disorder (MDD) or depressive episode of bipolar disorder (Bipolar I, II or NOS)
* Depression severity as defined by score of < 12 on the 21-item Hamilton Rating Scale for Depression and no psychiatric admission within 6 months from study entry and no suicide attempt within the last 12 months
* Willingness to sign human subjects consent form

Exclusion Criteria:

* Diagnosis of possible or probable cognitive impairment
* For women only: pregnancy, breastfeeding
* Personal history of Type I or Type II diabetes
* Unstable cardiovascular disease or other major medical condition, or history of myocardial infarction within the previous year
* Significant cerebrovascular disease, as evidenced by neurological examination, uncontrolled hypertension (systolic blood pressure > 170 or diastolic blood pressures > 100)
* Current drug or alcohol abuse
* History of neurological disorder, e.g. multiple sclerosis, stroke etc
* Use of any drug that may significantly affect psychometric testing or the insulin testing

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-11; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Rasgon, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Department of Psychiatry & Behavioral Sciences, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rasgon N, Lin KW, Lin J, Epel E, Blackburn E. Telomere length as a predictor of response to Pioglitazone in patients with unremitted depression: a preliminary study. Transl Psychiatry. 2016 Jan 5;6(1):e709. doi: 10.1038/tp.2015.187. PMID 26731446

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pioglitazone | Sugar Pill
Started | 19 | 18
Completed | 19 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | Sugar Pill | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 37
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.42 (15.11) | 43.28 (11.80) | 46.35 (13.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale at Baseline
Description: The HDRS-21 was used to screen for unremitted depression. The HDRS-21 is scored on a scale from 0 to 21, where 0 is the lowest level of depression severity and 21 is the highest level of depression severity. Unremitted depression is characterized by a score of ≥7. The HDRS-21 scores at baseline are shown in the data table below.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pio - IS: Participants who received pioglitazone and were insulin sensitive.
- Placebo - IS: Participants who received placebo and were insulin sensitive.
- Pio - IR: Participants who received pioglitazone and were insulin resistant.
- Placebo - IR: Participants who received the sugar pill and were insulin resistant.
Arm/Group | Pio - IS | Placebo - IS | Pio - IR | Placebo - IR
Number analyzed (Participants) | 9 | 8 | 10 | 10
units on a scale | 15.22 (2.64) | 13.67 (1.51) | 19.22 (7.26) | 13.25 (4.91)

2. Secondary Outcome: Fasting Insulin Measurements at Baseline
Description: The fasting plasma insulin measurements taken at baseline are shown in the data table below.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: uIU/mL
Arm/Group | Pio - IS | Placebo - IS | Pio - IR | Placebo - IR
Number analyzed (Participants) | 9 | 8 | 10 | 10
uIU/mL | 10.61 (2.49) | 9.18 (3.98) | 13.98 (6.35) | 14.12 (4.42)

3. Secondary Outcome: Change in HDRS-21: From Baseline to 12 Weeks
Description: The HDRS-21 was administered at baseline and at the end of 12 weeks, and the mean difference between the two time points was calculated. The HDRS-21 is scored on a scale from 0 to 21, where 0 is the lowest level of depression severity and 21 is the highest level of depression severity.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pio - IS | Placebo - IS | Pio - IR | Placebo - IR
Number analyzed (Participants) | 9 | 8 | 10 | 10
units on a scale | -4.45 (2.34) | -3.57 (1.9) | -1.71 (3.55) | -3.57 (5.77)

ADVERSE EVENTS:
Time Frame: The study period was 12 weeks.
Arm/Group | Pioglitazone | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No